CLINICAL TRIAL: NCT00041132
Title: Pilot Trial of Hyper-CVAD and Methotrexate/ARA C Plus Rituximab in Patients With Previously Untreated Mantle Cell Lymphoma
Brief Title: S0213 Chemotherapy Plus Rituximab in Treating Patients With Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069445; U10CA032102 (NIH); S0213 (Other: SWOG)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Results first posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Lymphoma
Keywords: stage III mantle cell lymphoma; stage IV mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Rituximab; Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Leucovorin; Methotrexate; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyper-CVAD + MTX/Ara-C + Rituximab (Experimental): 21-day cycles of Hyper-CVAD and high-dose methotrexate/cytarabine are alternated beginning with Hyper-CVAD for a maximum of 8 cycles. Rituximab is given for cycles 1-6.
  Hyper-CVAD (cycles 1,3,5,7): rituximab 375 mg/m^2 on day 1, mesna 600 mg/m^2 on days 2-4, cyclophosphamide 300 mg/m^2 on days 2-4, doxorubicin 16.6 mg/m^2/day on days 5-7, vincristine 1.4 mg/m^2 on days 5 and 12, dexamethasone 40 mg on days 2-5 and 12-15, and filgrastim 5 ug/kg on days 8-21.
  Methotrexate/Ara-C (cycles 2,4,6,8): rituximab 375 mg/m^2 on day 1, methotrexate 1000 mg/m^2 over days 2-3, Ara-C 12 g/m^2 over days 3-4, leucovorin 170 mg over days 3-5, and G-CSF 5 ug/kg on days 5-21.
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexamethasone; Drug: doxorubicin; Drug: leucovorin; Drug: methotrexate; Drug: vincristine

INTERVENTIONS:
Biological: filgrastim — 5 ug/kg
  Other Names: G-CSF
Biological: rituximab — 375 mg/m^2 on day 1 of cycles 1-6
Drug: cyclophosphamide — 300 mg/m^2 on days 2-4 of cycles 1,3,5,7
  Other Names: cytoxan
Drug: cytarabine — 12 g/m^2 over days 3-4 of cycles 2,4,6,8
  Other Names: Ara-C
Drug: dexamethasone — 40 mg on days 2-5 and 12-15 of cycles 1,3,5,7
Drug: doxorubicin — 16.6 mg/m^2/day for days 5-7 of cycles 1,3,5,7
  Other Names: adriamycin
Drug: leucovorin — 170 mg over days 3-5 of cycles 2,4,6,8
  Other Names: leucovorin calcium
Drug: methotrexate — 1000 mg/m^2 over days 2-3 of cycles 2,4,6,8
  Other Names: MTX
Drug: vincristine — 1.4 mg/m^2 on days 5 and 12 of cycles 1,3,5,7
  Other Names: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining rituximab with chemotherapy may kill more cancer cells.

PURPOSE: Phase II pilot study to study the effectiveness of combining chemotherapy with rituximab in treating patients who have newly diagnosed mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 1-year progression-free survival probability in patients with previously untreated mantle cell lymphoma treated with courses of rituximab and cyclophosphamide, doxorubicin, vincristine, and dexamethasone alternating with courses of rituximab and high-dose cytarabine and methotrexate with leucovorin calcium.
* Determine the response rate (complete unconfirmed and complete and partial responses) and survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Correlate chromosomal breakpoints, translocated immunoglobulin regulatory sequences, and cyclins D1, D2, and D3 with response and progression-free survival in patients treated with this regimen.
* Correlate gene expression (measured by DNA microarray analysis) with response and progression-free survival in patients treated with this regimen.

OUTLINE: This is a pilot, multicenter study.

* Courses 1, 3, 5, and 7: Patients receive rituximab IV on day 1 (courses 1, 3, and 5 only); cyclophosphamide IV over 3 hours twice a day on days 2-4; doxorubicin IV over 24 hours on days 5-7; vincristine IV on days 5 and 12; dexamethasone orally or IV four times a day on days 2-5 and 12-15; and filgrastim (G-CSF) subcutaneously (SC) daily beginning on day 8 and continuing until blood counts recover.
* Courses 2, 4, 6, and 8: Patients receive rituximab IV on day 1 (courses 2, 4, and 6 only); high-dose methotrexate IV over 24 hours on day 2; high-dose cytarabine IV over 2 hours twice a day on days 3-4; oral leucovorin calcium 4 times a day on days 3-10; and G-CSF SC daily beginning on day 5 and continuing until blood counts recover.

Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed within 30 days, every 3 months for 2 years, and then every 6 months for 3 years. Patients with disease progression are followed annually for up to 5 years from study entry.

PROJECTED ACCRUAL: Approximately 50 patients will be accrued for this study within 25 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage III/IV or bulky stage II mantle cell lymphoma of one of the following histologic subtypes:

  * Nodular
  * Diffuse
  * Mantle zone
  * Blastic
* Newly diagnosed and previously untreated disease
* Bidimensionally measurable disease

PATIENT CHARACTERISTICS:

Age:

* 18 to 69

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3 (50,000/mm^3 if marrow involvement present)

Hepatic:

* Bilirubin no greater than 1.5 mg/dL (5.0 mg/dL if hepatic involvement present)

Renal:

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance greater than 50 mL/min

Cardiovascular:

* Ejection fraction at least 50% by MUGA or 2-D echocardiogram
* No significant abnormalities by EKG

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Willing to receive blood product transfusions
* No known sensitivity to E. coli-derived proteins
* No known AIDS syndrome or HIV-associated complex
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior monoclonal antibody therapy

Chemotherapy:

* No prior chemotherapy for lymphoma

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for lymphoma

Surgery:

* Not specified

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2002-09; Primary Completion 2007-11 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot M. Epner, MD, PhD, Study Chair — OHSU Knight Cancer Institute

REFERENCES:
- [Result] A multi center trial of hyperCVAD+rituxan in patients with newly diagnosed mantle cell lymphoma EM Epner; J Unger; T Miller; L Rimsza; C Spier; M LeBlanc; R Fisher. Blood 110(11):#387. (2007).

RESULTS

PARTICIPANT FLOW:
Groups:
- Hyper-CVAD + MTX/Ara-C + Rituximab: 21-day cycles of Hyper-CVAD and high-dose methotrexate/Ara-C are alternated beginning with Hyper-CVAD for a maximum of 8 cycles. Rituximab is given for cycles 1-6.
  Hyper-CVAD (cycles 1,3,5,7): rituximab 375 mg/m^2 on day 1, mesna 600 mg/m^2 on days 2-4, cyclophosphamide 300 mg/m^2 on days 2-4, doxorubicin 16.6 mg/m^2/day on days 5-7, vincristine 1.4 mg/m^2 on days 5 and 12, dexamethasone 40 mg on days 2-5 and 12-15, and G-CSF 5 ug/kg on days 8-21.
  Methotrexate/Ara-C (cycles 2,4,6,8): rituximab 375 mg/m^2 on day 1, methotrexate 1000 mg/m^2 over days 2-3, Ara-C 12 g/m^2 over days 3-4, leucovorin 170 mg over days 3-5, and G-CSF 5 ug/kg on days 5-21.
Period: Overall Study
Arm/Group | Hyper-CVAD + MTX/Ara-C + Rituximab
Started | 56
Eligible | 49
Eligible and Began Protocol Therapy | 49
Completed | 26
Not Completed | 30
Not completed — Adverse Event | 19
Not completed — Death | 1
Not completed — Not Eligible | 7
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hyper-CVAD + MTX/Ara-C + Rituximab
Number analyzed (Participants) | 49
Age Continuous [Median (Full Range); unit: years] | 57.4 [35.0 to 69.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-Free Survival (PFS) rate at 1 year. PFS measured from date of registration to date of first observation of progressive disease or death due to any cause. Progressive disease is a 50% increase in the sum of products of greatest diameters (SPD) of target measurable lesions over the smallest sum observed if a complete response (confirmed, or unconfirmed) was not previously achieved; appearance of a new lesion/site; unequivocal progression of non-measurable disease; or death due to disease without prior documentation of progression.
Time Frame: assessed after cycle 4, after completion of treatment, then every 3 months until 1 year after registration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hyper-CVAD + MTX/Ara-C + Rituximab
Number analyzed (Participants) | 49
percentage of participants | 90 [77 to 96]

2. Secondary Outcome: Response
Description: Complete (CR), complete unconfirmed (CRU) and partial responses (PR). CR is complete disappearance of all measurable and non-measurable disease with the exception of nodes; no new lesions; previously enlarged organs must have regressed in size; and if bone marrow positive at baseline, it must be negative. CRU is complete disappearance of all measurable and non-measurable disease; regressed, non-palpable organs; and one or more exceptions not qualifying for CR (see protocol section 10). PR applies to patients with at least one measurable lesion who do not qualify for CR or CRU. PR is a 50% decrease in sum of products of greatest diameters (SPD) for up to six identified dominant lesions identified at baseline; no new lesions; no increase in the size of liver, spleen or other nodes; and splenic and hepatic nodules must have regressed in size by at least 50% in SPD.
Time Frame: assessed after cycle 4 and after completion of treatment (168 days)
Measure: Number; unit: participants
Arm/Group | Hyper-CVAD + MTX/Ara-C + Rituximab
Number analyzed (Participants) | 49
participants | 42

3. Secondary Outcome: Overall Survival
Description: Overall Survival rate at 1 year. Time to death is from date of registration to date of death due to any cause.
Time Frame: assessed after cycle 4, after completion of treatment, then every 3 months for 2 years, then every 6 months thereafter until 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hyper-CVAD + MTX/Ara-C + Rituximab
Number analyzed (Participants) | 49
percentage of participants | 92 [79 to 97]

ADVERSE EVENTS:
Time Frame: Every week while on protocol treatment (through 8 cycles or 168 days), and 3 months after removal from protocol treatment (at between 8 and 9 months after beginning treatment).
Arm/Group | Hyper-CVAD + MTX/Ara-C + Rituximab
Serious Adverse Events (participants affected / at risk) | 4/49
Other Adverse Events (participants affected / at risk) | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hyper-CVAD + MTX/Ara-C + Rituximab (N=49)
Colitis (Gastrointestinal disorders) | 1
Infection with 3-4 neutropenia (Infections and infestations) | 1
Second primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (incoordination) (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hyper-CVAD + MTX/Ara-C + Rituximab (N=49)
Anemia (Blood and lymphatic system disorders) | 45
Febrile neutropenia (Blood and lymphatic system disorders) | 10
PRBC transfusion (Blood and lymphatic system disorders) | 12
Platelet transfusion (Blood and lymphatic system disorders) | 8
Sinus tachycardia (Cardiac disorders) | 5
Blurred vision (Eye disorders) | 4
Dry eye (Eye disorders) | 3
Abdominal pain/cramping (Gastrointestinal disorders) | 3
Constipation/bowel obstruction (Gastrointestinal disorders) | 23
Diarrhea without colostomy (Gastrointestinal disorders) | 17
Dyspepsia/heartburn (Gastrointestinal disorders) | 4
Esophagitis/dysphagia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 20
Stomatitis/pharyngitis (Gastrointestinal disorders) | 26
Vomiting (Gastrointestinal disorders) | 15
Edema (General disorders) | 23
Fatigue/malaise/lethargy (General disorders) | 43
Fever without neutropenia (General disorders) | 20
Hemorrhage w/ 3-4 thrombocyt (General disorders) | 5
Pain-other (General disorders) | 3
Rigors/chills (General disorders) | 8
Allergic reaction (Immune system disorders) | 5
Infection w/o 3-4 neutropenia (Infections and infestations) | 15
Infection with 3-4 neutropenia (Infections and infestations) | 15
Respiratory infect w/ neutrop (Infections and infestations) | 3
Respiratory infect w/o neutrop (Infections and infestations) | 4
Alkaline phosphatase increase (Investigations) | 8
Bilirubin increase (Investigations) | 7
Creatinine increase (Investigations) | 6
Leukopenia (Investigations) | 44
Lymphopenia (Investigations) | 31
Neutropenia/granulocytopenia (Investigations) | 45
SGOT (AST) increase (Investigations) | 18
SGPT (ALT) increase (Investigations) | 10
Thrombocytopenia (Investigations) | 43
Anorexia (Metabolism and nutrition disorders) | 9
Hyperglycemia (Metabolism and nutrition disorders) | 22
Hyperuricemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 13
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 15
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 9
Muscle weakness (not neuro) (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Myalgia/arthralgia, NOS (Musculoskeletal and connective tissue disorders) | 3
Ataxia (incoordination) (Nervous system disorders) | 4
Dizziness/vertigo, NOS (Nervous system disorders) | 7
Headache (Nervous system disorders) | 17
Sensory neuropathy (Nervous system disorders) | 26
Taste disturbance (Nervous system disorders) | 3
Anxiety/agitation (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 7
Urinary frequency/urgency (Renal and urinary disorders) | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 35
Dry skin (Skin and subcutaneous tissue disorders) | 3
Petechiae/purpura (Skin and subcutaneous tissue disorders) | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 16
Hypotension (Vascular disorders) | 10
Phlebitis (Vascular disorders) | 3
Thrombosis/embolism (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No